CLINICAL TRIAL: NCT00195858
Title: Healthy Eating, Aerobic and Resistance Training in Youth (HEARTY) Trial
Brief Title: Healthy Eating Aerobic and Resistance Training in Youth (HEARTY) Trial
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Canadian Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: MCT-71979
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Obesity
Keywords: Youth; Exercise; Physical Activity; Aerobic; Resistance; Overweight; obese; Canada; Sigal
MeSH Terms: conditions — Obesity; Motor Activity; Overweight

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Diet and Aerobic Exercise (Active Comparator)
  Interventions: Behavioral: aerobic and resistance exercise
- Diet and Resistane Exercise (Active Comparator)
  Interventions: Behavioral: aerobic and resistance exercise
- Diet and Combined Aerobic and Resistance Exercise (Active Comparator)
  Interventions: Behavioral: aerobic and resistance exercise
- Diet-only control group (Other)
  Interventions: Behavioral: aerobic and resistance exercise

INTERVENTIONS:
Behavioral: aerobic and resistance exercise — aerobic and resistance exercise
  Other Names: non applicable

SUMMARY:
The purpose of this study is to evaluate the effects of resistance training, aerobic training, and combined aerobic and resistance training on percent body fat, measured using Magnetic Resonance Imaging (MRI), in sedentary post-pubertal overweight or obese youth aged 14-18 years.

DETAILED DESCRIPTION:
Background: Obesity and inactivity independently increase risks of chronic disease in adolescence and all-cause mortality in adulthood. In clinical trials, changes in exercise and diet can reduce adiposity and risk of diabetes and other chronic diseases in obese adults and youth. In many school systems, physical education is mandatory in elementary school but not high school, and physical activity often declines during adolescence. Because physical activity habits track from adolescence to adulthood, adolescence may represent a critical period for establishing a physically active lifestyle to prevent diseases associated with inactivity in adulthood. Obesity can make adherence to aerobic activity challenging, but would present less of an obstacle to resistance training. Resistance exercise has shown favorable effects on lean body mass, metabolic rate, insulin resistance, and quality of life in adults, but almost no research has examined effects of resistance training in obese adolescents. Our own survey in a sample of obese, primarily sedentary youth found greater overall interest in resistance exercise than aerobic exercise.

Objectives: The primary objective of this study is to evaluate the effects of resistance training, aerobic training, and combined aerobic and resistance training on percent body fat measured using Magnetic Resonance Imaging (MRI) in sedentary post-pubertal overweight or obese youth aged 14-18 years.

Study Design: Randomized controlled trial conducted at a single site. After a 4-week supervised low-intensity exercise run-in period to test compliance, 292 adolescents with BMI ≥ 85th percentile for age and gender will be randomized in equal numbers to one of 4 arms: Diet + aerobic exercise, diet + resistance exercise, diet + combined aerobic and resistance exercise, or diet-only control. The intervention will last 22 weeks, with a follow-up assessment at 6-months post-treatment (11-months post-randomization).

Hypotheses: Reduction in percent body fat will be larger in diet + aerobic exercise and diet + resistance exercise than diet-only controls at post-treatment, and the combined aerobic and resistance training will be superior to either aerobic or resistance training alone in reducing percent body fat at post-treatment. The combined resistance and aerobic group will show greater improvements in percent body fat, body composition, and physiological and psychosocial function at post-treatment and 12-months follow-up. Groups that include resistance training will produce greater psychosocial changes and better adherence than aerobic training alone at post-treatment and follow-up.

Significance: The global burden of obesity in youth is increasing, and more effective intervention is needed. This study may identify that resistance training is an important component in the treatment of overweight adolescents. As such, findings may influence clinical decision making in the management of juvenile obesity, as well as inform public health exercise guidelines and school-based physical education curricula in attempt to reduce the economic, medical, and psychosocial burden of obesity in youth.

ELIGIBILITY:
Inclusion Criteria:

* Male or female;
* aged 14-18 years,
* Tanner stage IV or above,
* waist circumference ≥75th percentile for age/gender
* body mass index ≥95th percentile for age, and gender
* AND/OR ≥85th percentile for age/gender with any of:
* Fasting glucose ≥6.0 fasting,
* 2-hour plasma glucose 7.8-11 mmol/L after 75 G oral glucose,
* fasting triglycerides > 1.7 mmol/L,
* fasting plasma insulin >105 pmol/L,
* HDL-C<0.9 mmol/L, LDL-C>3.0 mmol/L,
* total cholesterol/HDL-C >90th percentile,
* or first-degree relative with type 2 diabetes

Exclusion Criteria:

* Participation during the previous 4 months in a regular program of exercise or aerobic sports greater than 2 times per week for at least 20 minutes per session.
* Diabetes mellitus.
* Body weight over 159 kg, and/or BMI>45 kg/m2, exceeding capacity of DEXA and CT machines.
* Use of any performance-enhancing medication.
* Use of any medication or herbal supplement that is likely to affect body composition, lipids or glucose metabolism.
* Significant weight change (increase of ≥10%, or decrease≥5% of body weight during the two months before enrollment).
* Uncontrolled hypertension: BP >150 mm Hg systolic or >95 mm Hg diastolic BP in sitting position.
* Activity restrictions due to disease: unstable cardiac or pulmonary disease, significant arthritis.
* Other illness judged by the patient or study physician to make participation in this study inadvisable.
* Unwillingness/lack of availability to attend exercise and/or nutrition sessions at scheduled times and locations.
* Significant cognitive deficit resulting in inability to understand or comply with instructions.
* Pregnancy at the start of the study, or intention to become pregnant in the next year.
* Inability to communicate in English or French.
* Unwillingness of subject and/or parent/guardian to sign informed consent.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 304 (Actual)
Dates: Start 2005-04; Primary Completion 2010-11 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
change in percent body fat (MRI scan) | end of study

SECONDARY OUTCOMES:
Resting energy expenditure (indirect calorimetry). | end of study
Lean body mass | end of study
abdominal visceral and subcutaneous fat | end of study
waist and hip circumference | end of study
Apolipoprotein A1 | end of study
plasma insulin | end of study
HOMA insulin resistance | end of study
apoprotein B | end of study
C-reactive protein | end of study
HDL-C | end of study
LDL-C | end of study
triglycerides | end of study
total/HDL cholesterol ratio | end of study
fasting and 2-hour postload glucose | end of study
HbA1c | end of study
BP | end of study
Health related quality of life | end of study

CONTACTS AND LOCATIONS:
Overall Officials: Ronald J Sigal, MD MPH FRCPC, Principal Investigator — Ottawa Hospital Research Institute, University of Ottawa and the Ottawa Hospital
Locations (1):
- Ottawa Hospital Research Institute, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Alberga AS, Edache IY, Sigal RJ, von Ranson KM, Russell-Mayhew S, Kenny GP, Doucette S, Prud'homme D, Hadjiyannakis S, Cameron JD, Goldfield GS. Effects of the HEARTY exercise randomized controlled trial on eating behaviors in adolescents with obesity. Obes Sci Pract. 2022 Sep 6;9(2):158-171. doi: 10.1002/osp4.620. eCollection 2023 Apr. PMID 37034563
- [Derived] Goldfield GS, Walsh J, Sigal RJ, Kenny GP, Hadjiyannakis S, De Lisio M, Ngu M, Prud'homme D, Alberga AS, Doucette S, Goldfield DB, Cameron JD. Associations of the BDNF Val66Met Polymorphism With Body Composition, Cardiometabolic Risk Factors, and Energy Intake in Youth With Obesity: Findings From the HEARTY Study. Front Neurosci. 2021 Nov 12;15:715330. doi: 10.3389/fnins.2021.715330. eCollection 2021. PMID 34867148
- [Derived] Goldfield GS, Cameron JD, Sigal RJ, Kenny GP, Holcik M, Prud'homme D, Guerin E, Alberga AS, D'Angiulli A, Tremblay MS, Mougharbel F, Walsh J. Screen time is independently associated with serum brain-derived neurotrophic factor (BDNF) in youth with obesity. Appl Physiol Nutr Metab. 2021 Sep;46(9):1083-1090. doi: 10.1139/apnm-2020-0756. Epub 2021 Apr 8. PMID 33829867
- [Derived] Walsh JJ, D'Angiulli A, Cameron JD, Sigal RJ, Kenny GP, Holcik M, Doucette S, Alberga AS, Prud'homme D, Hadjiyannakis S, Gunnell K, Goldfield GS. Changes in the Brain-Derived Neurotrophic Factor Are Associated with Improvements in Diabetes Risk Factors after Exercise Training in Adolescents with Obesity: The HEARTY Randomized Controlled Trial. Neural Plast. 2018 Sep 30;2018:7169583. doi: 10.1155/2018/7169583. eCollection 2018. PMID 30363954
- [Derived] Goldfield GS, Kenny GP, Prud'homme D, Holcik M, Alberga AS, Fahnestock M, Cameron JD, Doucette S, Hadjiyannakis S, Tulloch H, Tremblay MS, Walsh J, Guerin E, Gunnell KE, D'Angiulli A, Sigal RJ. Effects of aerobic training, resistance training, or both on brain-derived neurotrophic factor in adolescents with obesity: The hearty randomized controlled trial. Physiol Behav. 2018 Jul 1;191:138-145. doi: 10.1016/j.physbeh.2018.04.026. Epub 2018 Apr 19. PMID 29679660
- [Derived] Cameron JD, Maras D, Sigal RJ, Kenny GP, Borghese MM, Chaput JP, Alberga AS, Goldfield GS. The mediating role of energy intake on the relationship between screen time behaviour and body mass index in adolescents with obesity: The HEARTY study. Appetite. 2016 Dec 1;107:437-444. doi: 10.1016/j.appet.2016.08.101. Epub 2016 Aug 18. PMID 27545672
- [Derived] Goldfield GS, Kenny GP, Alberga AS, Prud'homme D, Hadjiyannakis S, Gougeon R, Phillips P, Tulloch H, Malcolm J, Doucette S, Wells GA, Ma J, Cameron JD, Sigal RJ. Effects of aerobic training, resistance training, or both on psychological health in adolescents with obesity: The HEARTY randomized controlled trial. J Consult Clin Psychol. 2015 Dec;83(6):1123-35. doi: 10.1037/ccp0000038. Epub 2015 Aug 31. PMID 26322787
- [Derived] Alberga AS, Prud'homme D, Kenny GP, Goldfield GS, Hadjiyannakis S, Gougeon R, Phillips P, Malcolm J, Wells G, Doucette S, Ma J, Sigal RJ. Effects of aerobic and resistance training on abdominal fat, apolipoproteins and high-sensitivity C-reactive protein in adolescents with obesity: the HEARTY randomized clinical trial. Int J Obes (Lond). 2015 Oct;39(10):1494-500. doi: 10.1038/ijo.2015.133. Epub 2015 Jul 23. PMID 26202452
- [Derived] Goldfield GS, Cameron JD, Murray M, Maras D, Wilson AL, Phillips P, Kenny GP, Hadjiyannakis S, Alberga AS, Tulloch H, Doucette S, Sigal RJ. Screen time is independently associated with health-related quality of life in overweight and obese adolescents. Acta Paediatr. 2015 Oct;104(10):e448-54. doi: 10.1111/apa.13073. Epub 2015 Jul 14. PMID 26096064
- [Derived] Sigal RJ, Alberga AS, Goldfield GS, Prud'homme D, Hadjiyannakis S, Gougeon R, Phillips P, Tulloch H, Malcolm J, Doucette S, Wells GA, Ma J, Kenny GP. Effects of aerobic training, resistance training, or both on percentage body fat and cardiometabolic risk markers in obese adolescents: the healthy eating aerobic and resistance training in youth randomized clinical trial. JAMA Pediatr. 2014 Nov;168(11):1006-14. doi: 10.1001/jamapediatrics.2014.1392. PMID 25243536
- [Derived] Goldfield GS, Saunders TJ, Kenny GP, Hadjiyannakis S, Phillips P, Alberga AS, Tremblay MS, Sigal RJ. Screen viewing and diabetes risk factors in overweight and obese adolescents. Am J Prev Med. 2013 Apr;44(4 Suppl 4):S364-70. doi: 10.1016/j.amepre.2012.11.040. PMID 23498300
- [Derived] Alberga AS, Goldfield GS, Kenny GP, Hadjiyannakis S, Phillips P, Prud'homme D, Tulloch H, Gougeon R, Wells GA, Sigal RJ. Healthy Eating, Aerobic and Resistance Training in Youth (HEARTY): study rationale, design and methods. Contemp Clin Trials. 2012 Jul;33(4):839-47. doi: 10.1016/j.cct.2012.04.004. Epub 2012 Apr 21. PMID 22548962
- [Derived] Goldfield GS, Kenny GP, Hadjiyannakis S, Phillips P, Alberga AS, Saunders TJ, Tremblay MS, Malcolm J, Prud'homme D, Gougeon R, Sigal RJ. Video game playing is independently associated with blood pressure and lipids in overweight and obese adolescents. PLoS One. 2011;6(11):e26643. doi: 10.1371/journal.pone.0026643. Epub 2011 Nov 1. PMID 22069461
- See also: Related Info — http://www.ohri.ca